CLINICAL TRIAL: NCT04962087
Title: Randomized Controlled Trial to Evaluate Health enSuite Insomnia: an App-based Treatment for Adult Chronic Insomnia
Brief Title: Health enSuite Insomnia: an App-based Treatment for Adult Chronic Insomnia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Patrick J. McGrath, Principal Investigator, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1026706
Record Dates: First submitted 2021-06-14; First posted 2021-07-14 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Insomnia
Keywords: Insomnia; Deprescribing; Cognitive Behavioural Therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This project consists of a pragmatic randomized controlled trial (RCT). The Consolidated Standards of Reporting Trials (CONSORT) recommendations (http://www.consort-statement.org/) will guide the methodology. Participants will be randomly allocated in a 1:1 ratio to either the intervention group or a waitlist control group.
  Participants in both groups will complete self-assessments including key outcome measures at baseline before starting the study, at two months post-randomization, and again at five months post-randomization. Participants in the intervention group will receive the full Health enSuite Insomnia program immediately after being randomized to this group. Participants in the waitlist control group will be waitlisted during the study. After their participation in the study has ended, participants in the waitlist control group will be given access to the full Health enSuite Insomnia program for two months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health enSuite Insomnia (Experimental): Health enSuite: Insomnia has been designed based on established cognitive behavioral treatments for insomnia (2,5,6) and adapted to fit an automated interactive platform available via an internet enabled device. Previous research has found that CBT for insomnia can be delivered via a web-based platform (15,16). The program is divided into a series of treatment modules or levels that will be delivered over the course of 8 weeks. The content of these 8 levels includes the following components, a sleep diary, Introduction to Health EnSuite Insomnia, Sleep restriction clock, Medications, Herbal Remedies & Sleep, Chronobiology & Sleep Timing, Sleep hygiene, Relaxation techniques, Changing Negative Thoughts Related to Sleep, Light and Sleep.
  Interventions: Behavioral: Experimental: Health enSuite Insomnia
- Waitlist Control (No Intervention): Participants allocated to the control group will not have access to Health enSuite Insomnia CBT-I content until the end of the trial. During the trial, they will receive treatment as usual and will not be restricted from accessing other standard care services for insomnia treatment.

INTERVENTIONS:
Behavioral: Experimental: Health enSuite Insomnia — Health enSuite: Insomnia has been designed based on established cognitive behavioral treatments for insomnia (2,5,6) and adapted to fit an automated interactive platform available via an internet enabled device. Previous research has found that CBT for insomnia can be delivered via a web-based platform (15,16). The program is divided into a series of treatment modules or levels that will be delivered over the course of 8 weeks. The content of these 8 levels includes the following components, a sleep diary, Introduction to Health EnSuite Insomnia, Sleep restriction clock, Medications, Herbal Remedies & Sleep, Chronobiology & Sleep Timing, Sleep hygiene, Relaxation techniques, Changing Negative Thoughts Related to Sleep, Light and Sleep.
  Arms: Health enSuite Insomnia

SUMMARY:
This project consists of a randomized controlled trial. The objective of this trial is to test the effectiveness of an app-based cognitive behavioral program for insomnia (Health enSuite: Insomnia) in reducing insomnia symptoms.

DETAILED DESCRIPTION:
Insomnia or insufficient sleep is one of the most prevalent public health issues. Nearly 1 in 4 Canadians over the age of 18 years report having difficulty falling asleep or maintaining sleep, the majority of whom have experienced these insomnia symptoms for more than a year. Chronic insomnia is characterized by one or more of the following symptoms occurring for at least three nights per week for at least 3 months: difficulty falling asleep, trouble maintaining sleep, difficulty in getting back to sleep, poor quality of sleep, and waking up too early the next morning. These symptoms persist despite adequate opportunity for sleep and are accompanied by significant impairments in daytime functioning.

Cognitive behavioral therapy for insomnia (CBT-I) is a multi-component intervention approach that is recommended as the first line of treatment for patients with persistent insomnia. It targets beliefs, thoughts, and expectations related to sleep as well as behavioral factors that result in sleep loss (sleep schedules, caffeine intake prior to bedtime, bright light in bedroom). These interventions have been found to improve the quality and the duration of sleep and improve daytime functioning. Despite the efficacy of CBT-I programs, they are not readily available to most patients. Therefore, our goal is to develop a CBT-I program that can be delivered through an internet connected phone, tablet, or computer and provide effective treatment to a wide range of people with chronic insomnia. Given that many individuals seek help for sleep problems online or face barriers accessing in-person care, internet-based CBT-I offers a scalable and accessible solution for those experiencing chronic insomnia.

Sleep medications are commonly used to manage insomnia symptoms. These include benzodiazepines such as temazepam and non-benzodiazepines like zopiclone, zolpidem, and zaleplon (often referred to as "Z drugs"). While these benzodiazepine receptor agonists (BZRAs) can be effective in the short term, long-term use is associated with diminishing benefits and potential risks, such as side effects, dependence, and-particularly in older adults-falls and cognitive impairment. Given these concerns, there is growing recognition of the importance of expanding access to non-pharmacological, evidence-based treatments for insomnia. Cognitive behavioral therapy for insomnia (CBT-I) is one such approach, but it remains underutilized due to limited availability. A widely accessible, app-based CBT-I program has the potential to fill this gap and offer a safer, long-term solution for individuals struggling with chronic insomnia.

This project consists of a randomized controlled trial. The objective of this trial is to test the effectiveness of an app-based cognitive behavioral program for insomnia (Health enSuite: Insomnia) in reducing insomnia symptoms.

The objectives will be to assess the effectiveness of CBT-I delivered through the Health enSuite app in:

* Reducing the severity of insomnia symptoms (primary outcome)
* Increasing sleep efficiency and total sleep time (secondary outcomes)
* Reducing sleep onset latency, time in bed, and the duration and frequency of awakenings at night (secondary outcomes)
* Reducing symptoms of psychological distress, anxiety, and depression (secondary outcomes) User engagement and satisfaction with Health enSuite: Insomnia will also be evaluated to inform subsequent efforts to make this program available on a larger scale.

ELIGIBILITY:
To be eligible for this study, participants must meet all of the following criteria:

* Age 18 years or older Rationale: The intervention is designed for adults. Sleep patterns, treatment needs, and legal capacity for consent differ in children and adolescents, so participants must be legal adults to provide informed consent and to ensure relevance of the treatment content.
* Experience one or more insomnia symptoms (e.g., difficulty falling asleep, staying asleep, or waking too early) at least 3 times per week for at least 3 months Rationale: This criterion aligns with standard diagnostic criteria for chronic insomnia (e.g., DSM-5, ICSD-3 (9,10), ensuring that the intervention targets individuals with persistent and clinically meaningful symptoms.
* Have access to an internet-connected device (e.g., smartphone, tablet, or computer) Rationale: The CBT-I program is delivered entirely online via a mobile app or web platform. Participants must have reliable access to an internet-enabled device to complete program content, questionnaires, and sleep diaries.
* Not currently working regular overnight shifts (e.g., shifts starting between 10:00 PM and 12:00 AM and ending between 6:00 AM and 8:00 AM) Rationale: Night shift work disrupts circadian rhythms and sleep patterns in ways that are distinct from chronic insomnia. Individuals who work night shifts may not benefit from a standardized sleep schedule and could face difficulties adhering to the intervention.
* Not currently a parent of an infant under 1 year of age Rationale: Caring for an infant often involves frequent nighttime awakenings and irregular sleep patterns that are not necessarily reflective of insomnia. These participants may be unable to maintain a consistent sleep schedule as required by the intervention.
* Not currently pregnant or trying to become pregnant. Rationale: Sleep disturbances during pregnancy often result from physiological and hormonal changes, which differ from behavioral insomnia. The program has not been designed or tested for use during pregnancy, and eligibility will change if pregnancy occurs during the study.
* Have a total score greater than 7 on the Insomnia Severity Index (ISI) (11), indicating at least mild insomnia symptoms.

Rationale: The ISI is a validated tool used to assess the severity of insomnia symptoms. A score of 8 or more indicates at least mild insomnia, which supports the need for intervention. Excluding participants with minimal or no symptoms ensures that the program is delivered to those who stand to benefit and that changes in symptoms are measurable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index (ISI) Score | Baseline assessment, 2 months post-randomization, 5 months post-randomization
  The ISI is a 7-item questionnaire measuring insomnia severity, dissatisfaction with sleep, interference with daily functioning, and daytime impairment. Scores range from 0-28, with higher scores indicating more severe insomnia.

SECONDARY OUTCOMES:
Change in Depression, Anxiety, and Stress Scores (DASS-21) | Baseline assessment, 2 months post-randomization, 5 months post-randomization
  The DASS-21 is a 21-item questionnaire measuring psychological distress across three subscales: depression, anxiety, and stress. Each item is scored 0-3, and higher scores indicate greater distress.
Change in Sleep Efficiency | Baseline assessment, 2 months post-randomization, 5 months post-randomization
  Sleep efficiency will be calculated from sleep diary data as the ratio of total sleep time to time in bed (percentage).
Change in Total Sleep Time | Baseline assessment, 2 months post-randomization, 5 months post-randomization
  Total sleep time in hours will be calculated from daily sleep diaries. Unit of Measure: Hours of sleep (hours/night).
Change in Sleep Onset Latency | Baseline assessment, 2 months post-randomization, 5 months post-randomization
  Sleep onset latency (minutes taken to fall asleep) will be measured via sleep diary.
  Unit of Measure: Minutes.
Change in Wake After Sleep Onset (WASO) | Baseline assessment, 2 months post-randomization, 5 months post-randomization
  WASO (total time awake after initially falling asleep) will be recorded via sleep diary.
  Unit of Measure: Minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick McGrath, Principal Investigator — IWK Health Centre
Locations (1):
- Centre for Research in Family Health, IWK Health, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified data sets may be retained and stored within the Centre for Research in Family Health as required for future research or program development, if merited. During Consent, participants will be offered the option of allowing their de-identified study data to be re-used by other approved researchers under the conditions that the research projects are approved by an appropriate ethics board and the researchers sign an agreement ensuring confidentiality and restricting data use only to the approved study. A database will be created containing only the data for those participants who agree will be available to researchers who meet these criteria.
Time Frame: From study closure to five years post publication.
Access Criteria: During Consent, participants will be offered the option of allowing their de-identified study data to be re-used by other approved researchers under the conditions that the research projects are approved by an appropriate ethics board and the researchers sign an agreement ensuring confidentiality and restricting data use only to the approved study. A database will be created containing only the data for those participants who agree will be available to researchers who meet these criteria.

REFERENCES:
- [Background] Chaput JP, Yau J, Rao DP, Morin CM. Prevalence of insomnia for Canadians aged 6 to 79. Health Rep. 2018 Dec 19;29(12):16-20. PMID 30566205
- [Background] Morin CM, Benca R. Chronic insomnia. Lancet. 2012 Mar 24;379(9821):1129-41. doi: 10.1016/S0140-6736(11)60750-2. Epub 2012 Jan 20. PMID 22265700
- [Background] Management of Chronic Insomnia Disorder in Adults: A Clinical Practice Guideline From the American College of Physicians. Ann Intern Med. 2016 Jul 19;165(2). doi: 10.7326/P16-9016. Epub 2016 May 3. No abstract available. PMID 27135191
- [Background] Schutte-Rodin S, Broch L, Buysse D, Dorsey C, Sateia M. Clinical guideline for the evaluation and management of chronic insomnia in adults. J Clin Sleep Med. 2008 Oct 15;4(5):487-504. PMID 18853708
- [Background] van Straten A, van der Zweerde T, Kleiboer A, Cuijpers P, Morin CM, Lancee J. Cognitive and behavioral therapies in the treatment of insomnia: A meta-analysis. Sleep Med Rev. 2018 Apr;38:3-16. doi: 10.1016/j.smrv.2017.02.001. Epub 2017 Feb 9. PMID 28392168
- [Background] Trauer JM, Qian MY, Doyle JS, Rajaratnam SM, Cunnington D. Cognitive Behavioral Therapy for Chronic Insomnia: A Systematic Review and Meta-analysis. Ann Intern Med. 2015 Aug 4;163(3):191-204. doi: 10.7326/M14-2841. PMID 26054060
- [Background] Koffel E, Bramoweth AD, Ulmer CS. Increasing access to and utilization of cognitive behavioral therapy for insomnia (CBT-I): a narrative review. J Gen Intern Med. 2018 Jun;33(6):955-962. doi: 10.1007/s11606-018-4390-1. Epub 2018 Apr 4. PMID 29619651
- [Background] Holbrook AM, Crowther R, Lotter A, Cheng C, King D. Meta-analysis of benzodiazepine use in the treatment of insomnia. CMAJ. 2000 Jan 25;162(2):225-33. PMID 10674059
- [Background] Pottie K, Thompson W, Davies S, Grenier J, Sadowski CA, Welch V, Holbrook A, Boyd C, Swenson R, Ma A, Farrell B. Deprescribing benzodiazepine receptor agonists: Evidence-based clinical practice guideline. Can Fam Physician. 2018 May;64(5):339-351. PMID 29760253
- [Background] Glass J, Lanctot KL, Herrmann N, Sproule BA, Busto UE. Sedative hypnotics in older people with insomnia: meta-analysis of risks and benefits. BMJ. 2005 Nov 19;331(7526):1169. doi: 10.1136/bmj.38623.768588.47. Epub 2005 Nov 11. PMID 16284208
- [Background] Farrell B, Tsang C, Raman-Wilms L, Irving H, Conklin J, Pottie K. What are priorities for deprescribing for elderly patients? Capturing the voice of practitioners: a modified delphi process. PLoS One. 2015 Apr 7;10(4):e0122246. doi: 10.1371/journal.pone.0122246. eCollection 2015. PMID 25849568
- [Background] Pollmann AS, Murphy AL, Bergman JC, Gardner DM. Deprescribing benzodiazepines and Z-drugs in community-dwelling adults: a scoping review. BMC Pharmacol Toxicol. 2015 Jul 4;16:19. doi: 10.1186/s40360-015-0019-8. PMID 26141716
- [Background] Lee JY, Farrell B, Holbrook AM. Deprescribing benzodiazepine receptor agonists taken for insomnia: a review and key messages from practice guidelines. Pol Arch Intern Med. 2019 Jan 31;129(1):43-49. doi: 10.20452/pamw.4391. Epub 2018 Dec 13. PMID 30543200
- [Background] Morin CM, Vallieres A, Guay B, Ivers H, Savard J, Merette C, Bastien C, Baillargeon L. Cognitive behavioral therapy, singly and combined with medication, for persistent insomnia: a randomized controlled trial. JAMA. 2009 May 20;301(19):2005-15. doi: 10.1001/jama.2009.682. PMID 19454639
- [Background] Ng BJ, Le Couteur DG, Hilmer SN. Deprescribing Benzodiazepines in Older Patients: Impact of Interventions Targeting Physicians, Pharmacists, and Patients. Drugs Aging. 2018 Jun;35(6):493-521. doi: 10.1007/s40266-018-0544-4. PMID 29705831
- [Background] Morin CM, LeBlanc M, Belanger L, Ivers H, Merette C, Savard J. Prevalence of insomnia and its treatment in Canada. Can J Psychiatry. 2011 Sep;56(9):540-8. doi: 10.1177/070674371105600905. PMID 21959029
- [Background] Zachariae R, Lyby MS, Ritterband LM, O'Toole MS. Efficacy of internet-delivered cognitive-behavioral therapy for insomnia - A systematic review and meta-analysis of randomized controlled trials. Sleep Med Rev. 2016 Dec;30:1-10. doi: 10.1016/j.smrv.2015.10.004. Epub 2015 Oct 24. PMID 26615572
- [Background] Cheung JMY, Jarrin DC, Ballot O, Bharwani AA, Morin CM. A systematic review of cognitive behavioral therapy for insomnia implemented in primary care and community settings. Sleep Med Rev. 2019 Apr;44:23-36. doi: 10.1016/j.smrv.2018.11.001. Epub 2018 Nov 23. PMID 30612061
- [Background] Ye YY, Zhang YF, Chen J, Liu J, Li XJ, Liu YZ, Lang Y, Lin L, Yang XJ, Jiang XJ. Internet-Based Cognitive Behavioral Therapy for Insomnia (ICBT-i) Improves Comorbid Anxiety and Depression-A Meta-Analysis of Randomized Controlled Trials. PLoS One. 2015 Nov 18;10(11):e0142258. doi: 10.1371/journal.pone.0142258. eCollection 2015. PMID 26581107
- [Background] Ritterband LM, Thorndike FP, Ingersoll KS, Lord HR, Gonder-Frederick L, Frederick C, Quigg MS, Cohn WF, Morin CM. Effect of a Web-Based Cognitive Behavior Therapy for Insomnia Intervention With 1-Year Follow-up: A Randomized Clinical Trial. JAMA Psychiatry. 2017 Jan 1;74(1):68-75. doi: 10.1001/jamapsychiatry.2016.3249. PMID 27902836
- [Background] Baillargeon L, Landreville P, Verreault R, Beauchemin JP, Gregoire JP, Morin CM. Discontinuation of benzodiazepines among older insomniac adults treated with cognitive-behavioural therapy combined with gradual tapering: a randomized trial. CMAJ. 2003 Nov 11;169(10):1015-20. PMID 14609970
- [Background] Voshaar RC, Gorgels WJ, Mol AJ, van Balkom AJ, van de Lisdonk EH, Breteler MH, van den Hoogen HJ, Zitman FG. Tapering off long-term benzodiazepine use with or without group cognitive-behavioural therapy: three-condition, randomised controlled trial. Br J Psychiatry. 2003 Jun;182:498-504. doi: 10.1192/bjp.182.6.498. PMID 12777340
- [Background] Olivier J, May WL, Bell ML. Relative effect sizes for measures of risk. Communications in Statistics-Theory and Methods 2017;46(14):6774-6781.
- [Background] Morin CM. Measuring outcomes in randomized clinical trials of insomnia treatments. Sleep Med Rev. 2003 Jun;7(3):263-79. doi: 10.1053/smrv.2002.0274. PMID 12927124
- [Background] Carney CE, Buysse DJ, Ancoli-Israel S, Edinger JD, Krystal AD, Lichstein KL, Morin CM. The consensus sleep diary: standardizing prospective sleep self-monitoring. Sleep. 2012 Feb 1;35(2):287-302. doi: 10.5665/sleep.1642. PMID 22294820
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Thorndike FP, Ritterband LM, Saylor DK, Magee JC, Gonder-Frederick LA, Morin CM. Validation of the insomnia severity index as a web-based measure. Behav Sleep Med. 2011;9(4):216-23. doi: 10.1080/15402002.2011.606766. PMID 22003975
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Antony MM, Bieling PJ, Cox BJ, Enns MW, Swinson RP. Psychometric properties of the 42-item and 21-item versions of the Depression Anxiety Stress Scales in clinical groups and a community sample. Psychol Assess 1998;10(2):176.
- [Background] Henry JD, Crawford JR. The short-form version of the Depression Anxiety Stress Scales (DASS-21): construct validity and normative data in a large non-clinical sample. Br J Clin Psychol. 2005 Jun;44(Pt 2):227-39. doi: 10.1348/014466505X29657. PMID 16004657
- [Background] Gloster AT, Rhoades HM, Novy D, Klotsche J, Senior A, Kunik M, Wilson N, Stanley MA. Psychometric properties of the Depression Anxiety and Stress Scale-21 in older primary care patients. J Affect Disord. 2008 Oct;110(3):248-59. doi: 10.1016/j.jad.2008.01.023. Epub 2008 Mar 4. PMID 18304648
- [Background] Attkisson CC, Greenfield TK. The UCSF Client Satisfaction Scales: I. The Client Satisfaction Questionnaire-8. In: Maruish ME, editor. The use of psychological testing for treatment planning and outcomes assessment: Instruments for adults Mahwah, NJ, US: Lawrence Erlbaum Associates Publishers; 2004. p. 799-799-811.
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Thorndike FP, Saylor DK, Bailey ET, Gonder-Frederick L, Morin CM, Ritterband LM. Development and Perceived Utility and Impact of an Internet Intervention for Insomnia. E J Appl Psychol. 2008;4(2):32-42. doi: 10.7790/ejap.v4i2.133. PMID 20953264
- [Background] Morin CM, Blais F, Savard J. Are changes in beliefs and attitudes about sleep related to sleep improvements in the treatment of insomnia? Behav Res Ther. 2002 Jul;40(7):741-52. doi: 10.1016/s0005-7967(01)00055-9. PMID 12074370
- [Background] Prochaska JO. Transtheoretical model of behavior change. Encyclopedia of behavioral medicine: Springer; 2013. p. 1997-2000.
- [Background] Rogojanski J, Carney CE, Monson CM. Interpersonal factors in insomnia: a model for integrating bed partners into cognitive behavioral therapy for insomnia. Sleep Med Rev. 2013 Feb;17(1):55-64. doi: 10.1016/j.smrv.2012.02.003. Epub 2012 May 18. PMID 22609123

DOCUMENTS (1):
  • Informed Consent Form (2024-02-26): https://cdn.clinicaltrials.gov/large-docs/87/NCT04962087/ICF_000.pdf